CLINICAL TRIAL: NCT03818113
Title: Clinical Comparative Analysis of Bretschneider and St. Thomas Cardioplegia Solution in Case of Mitral Valve Repair Via Anterolateral Right Thoracotomy
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-00070; ch18Grapow4
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Mitral Valve Reconstruction
Keywords: mitral valve insufficiency; cardioplegia; cardioplegia Solution; HTK-Bretschneider (Custidiol®) solution; St. Thomas solution; cardiac biomarker
MeSH Terms: conditions — Mitral Valve Insufficiency | interventions — Heart Arrest, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HTK-Bretschneider cardioplegic solution: Patients undergoing mitral valve reconstruction via minimal invasive antero- lateral thoracotomy in cardioplegia with HTK-Bretschneider cardioplegic solution
  Interventions: Other: cardioplegia with HTK-Bretschneider cardioplegic solution
- St. Thomas cardioplegic solution: Patients undergoing mitral valve reconstruction via minimal invasive antero- lateral thoracotomy in cardioplegia with St. Thomas cardioplegic solution
  Interventions: Other: cardioplegia with St. Thomas cardioplegic solution

INTERVENTIONS:
Other: cardioplegia with HTK-Bretschneider cardioplegic solution — cardioplegia with HTK-Bretschneider cardioplegic solution
  Groups: HTK-Bretschneider cardioplegic solution
Other: cardioplegia with St. Thomas cardioplegic solution — cardioplegia with St. Thomas cardioplegic solution
  Groups: St. Thomas cardioplegic solution

SUMMARY:
Mitral valve reconstruction via minimal invasive antero- lateral thoracotomy is done in cardioplegia with a cardioplegic solution, either HTK-Bretschneider (Custidiol®) (a crystalloid intracellular solution) or St. Thomas (a crystalloid extracellular solution).

This study investigates HTK-Bretschneider versus St. Thomas cardioplegic solution regarding peri- and postoperative outcome, especially for cardiac biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Mitral valve reconstruction via minimal invasive antero- lateral thoracotomy done in cardioplegia with a cardioplegic solution, either HTK-Bretschneider (Custidiol®) (a crystalloid intracellular solution) or St. Thomas (a crystalloid extracellular solution).

Exclusion Criteria:

* Mitral valve reconstruction via minimal invasive antero- lateral thoracotomy done in cardioplegia with cardioplegic Solutions other than HTK-Bretschneider (Custidiol®) (a crystalloid intracellular solution) or St. Thomas (a crystalloid extracellular solution).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with mitral valve reconstruction done via minimal invasive antero- lateral thoracotomy (2009-2018) at Universitätsspital Basel.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
high specific troponin T (hs-TrT) (μg/l) | perioperative during minimal invasive surgery
  cardial biomarker for myocardial damage
Creatin-Phosphokinase (CK) (U/l) | perioperative during minimal invasive surgery
  cardial biomarker for myocardial damage
Creatinkinase Muscle- Brain (CK-MB) (U/l) | perioperative during minimal invasive surgery
  cardial biomarker for myocardial damage

SECONDARY OUTCOMES:
mortality rate | from minimal invasive surgery until 30 days post surgery
  number of deaths
length of stay in intensive care unit (days) | from minimal invasive surgery until 30 days post surgery
  length of stay in intensive care unit (number of days)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grapow, Prof. Dr., Principal Investigator — Klinik für Herzchirurgie, Universitätsspital Basel
Locations (1):
- Klinik für Herzchirurgie, Universitätsspital Basel, Basel, Switzerland